CLINICAL TRIAL: NCT06798428
Title: Effect of Glucosamine, Chondroitin and Some Herbs Extract Phonophoresis in the Treatment of Grade I and II Knee Meniscal Injuries: a Randomized Placebo-controlled Clinical Trial.
Brief Title: For Grade I and II Knee Meniscal Injuries Patients ,Glucosamine, Chondroitin and Some Herbs Extract Phonophoresis Will Be Used (A) Versus Placebo(B)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eslam Elsayed Ali Shohda (Other Government)
Responsible Party: Sponsor-Investigator, Eslam Elsayed Ali Shohda, Dr Eslam Shohda-Principal Investigator, General Committee of Teaching Hospitals and Institutes, Egypt
Organization: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAH00014
Record Dates: First submitted 2025-01-11; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Grade I and II Knee Meniscal Injuries
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Massage

STUDY DESIGN:
Intervention Model Description: randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- expermental ( A) (Experimental): group A, will receive ultrasound phonophoresis (Glucosamine, Chondroitin and Some Herbs Extract ) Ultrasound parameters are 1 W/cm for intensity, 1 MHz for frequency and 5 min continuous mode then 5 min pulsed mode
  Interventions: Device: group A will receive ultrasound phonophoresis (Glucosamine, Chondroitin and Some Herbs Extract )
- B (Experimental): group B, will receive ultrasound with topical gel , same parameter as group A
  Interventions: Device: Group B will receive ultrasound with topical gel , same parameter as group A
- C (Sham Comparator): group C, will receive ultrasound( machine is off) massage for 5 minutes
  Interventions: Device: Group C sham ultrasound for massage - 5 minutes

INTERVENTIONS:
Device: group A will receive ultrasound phonophoresis (Glucosamine, Chondroitin and Some Herbs Extract ) — Group (A)will have GL, CH and natural herbs phonophoresis .Ultrasound parameters are 1 W/cm for intensity, 1 MHz for frequency and 5 min continuous mode then 5 min pulsed mode. The device that will be used is medserve, England (the head of the device is 5cm).
  Arms: expermental ( A)
Device: Group B will receive ultrasound with topical gel , same parameter as group A — Ultrasound parameters are 1 W/cm for intensity, 1 MHz for frequency and 5 min continuous mode then 5 min pulsed mode. The device that will be used is medserve, England (the head of the device is 5cm). Topical gel with no drugs
  Arms: B
Device: Group C sham ultrasound for massage - 5 minutes — sham ultrasound for massage - 5 minutes
  Arms: C

SUMMARY:
Hypothesis: In grade I and II meniscal injury patients, 1) GL and CH (PH) decrease knee pain severity measured by Numerical Rating Scales (NRS) more than only topical application. 2) GL and CH (PH) improve knee functional abilities measured by Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) more than only topical application.

DETAILED DESCRIPTION:
Design and Setting: We propose a randomized (1:1:1) controlled, clinical trial to enroll grade I and II knee meniscal injuries' patients and to study the effect of GL, CH and some natural herbs (PH) in decreasing knee pain intensity measured by NRS and improving knee functional abilities measured by WOMAC. The study will be conducted in physical therapy outpatient clinic at Alahrar teaching hospital, Zagazig, Egypt.

Inclusion and Exclusion criteria: patients will be included to this study

* if they have grade I or II knee meniscal tear assessed by MRI according to radiologist report
* positive McMurray's test assessed by physical therapist
* aged from 18 to 40 years.

Exclusion criteria:

* grade III meniscal injury as it is supposed that they need more physical therapy sessions.
* Ages above 40 is excluded to exclude arthritic changes.
* Presence of any other knee injury or systemic diseases affecting joints (e.g. rheumatoid arthritis) will be excluded.
* Patients with body mass index (BMI) more than 30 will be excluded as their knees may have some arthritic changes and need longer PT sessions.

Sample size calculation: By reviewing literature, it is found that the most relevant study (5) to this work found that the mean pain score for treatment group is 5.25 ± 1.90 and for control group is 6.67 ± 1.78 so, by using G power (3.1) to calculate sample size (power = 0.8, alpha error = 0.05 and beta= 0.2) it is found that we need 15 patients for every group (45 patients for 3 groups). It is suggested that this would take about 1 year to complete the study.

Procedures: Patients will be evaluated by same physical therapist (researcher) to check his/her eligibility to be included to the study. Randomized blocks will be used to insure 1:1:1 blocked randomization. Pain severity will be evaluated by using NRS. Patients will be asked to indicate his/her knee pain severity (while usual movement) on the scale (zero is minimum and 10 is maximum). Knee functional abilities will be measured by (WOMAC) questioner which assess knee through 3 main items: pain, stiffness and physical function. Age, weight and height will be recorded. Every patient will be assessed at the beginning of the study and after last sessions by 2 days. Group (A)will have GL, CH and natural herbs (PH); the patient will be at supine lying position with a small bellow under his knee, a 4 cm gel (GL and CH 5%) will be used while US insonation under the head of US. Duration of US application is 10 min.US parameters are 1 W/cm for intensity, 1 MHz for frequency and 5 min continuous mode then 5 min pulsed mode. The device that will be used is medserve, England (the head of the device is 5cm). Group (B) will have US insonation with the same parameters as group (A), but with US topical gel (no drug). Group (c) will have topical gel applied with the head of US (10 min) while the machine is switched off (applied as massage). All patients will be referred to PT outpatient clinic by the orthopedist that standardize the drug protocol (anti-inflammatory drug) for all refereed patients. The physical therapy will by 6 successive sessions weekly for 2 weeks (12 sessions). PT sessions will be done by the same physical therapist.

Ethical aspects:

All patients will have a good explanation of their disease and available treatment. All patients will be instructed about the study and they have the choice to participate or not. In all cases patients will have their treatment.

Analysis of results:

Age, weight, height and BMI are expressed by mean (M) and standard deviation(SD). ANOVA test will be used to test if there is significant difference between groups regarding these variables. Investigators will compare between the three groups regarding pain severity measured by NRS (ordinal variables) and functional abilities measured by WOMAC which are expressed as median and inter quartile range (M) (IQR) by using Kruskal-Wallis test. Investigators will use logistic regression to compare between groups regarding frequency of triggering. Differences will be considered significant at P <0.05. Confidence interval will be calculated at 95%. Regression analysis will be used to investigate possible confounders (Age, weight, height, BMI and sex) especially if there is significant difference between the two groups regarding age, BMI and sex.

ELIGIBILITY:
Inclusion Criteria:

* grade I or II knee meniscal tear assessed by MRI according to radiologist report, positive McMurray's test assessed by physical therapist and aged from 18 to 60 years.

Exclusion Criteria:

* We suggest not to include grade III meniscal injury as it is supposed that they need more physical therapy sessions. Ages above 40 is excluded to exclude arthritic changes. Presence of any other knee injury or systemic diseases affecting joints (e.g. rheumatoid arthritis) will be excluded. Patients with body mass index (BMI) more than 30 will be excluded as their knees may have some arthritic changes and need longer PT sessions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
pain severity measured by Numerical Rating Scales (NRS) | before intervention and two days after last session
  zero , no pain .10 maximum pain

SECONDARY OUTCOMES:
knee functional abilities measured by Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) | before intervention and two dayes after last sesssion
  Zero - no functional impairments.96 ,maximum impairments

CONTACTS AND LOCATIONS:
Locations (1):
- Al ahrar teaching hospital, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No